CLINICAL TRIAL: NCT00494637
Title: The Use of Sodium Bicarbonate in the Prevention of Contrast Induced Nephropathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not reaching recruitment and endpoint goals
Sponsor: Lenox Hill Hospital (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Jordan L. Rosenstock, MD, Lenox Hill Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: L06.10.058
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Contrast Induced Nephropathy
MeSH Terms: interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sodium bicarbonate — isotonic sodium bicarbonate at 3 cc/kg for one hour followed by 2 cc kg/hr for 4 hours

SUMMARY:
Preliminary studies have shown a benefit of sodium bicarbonate infusion in decreasing the risk of contrast induced nephropathy with coronary angiography. The investigators plan to randomize 478 patients (with serum creatinine 1.5 mg/dl or greater) undergoing coronary angiography to intravenous isotonic saline or intravenous isotonic sodium bicarbonate beginning one hour before the procedure and for four hours after. The primary endpoint is the development of contrast nephropathy within 48-72 hours after the procedure. Patients with an ejection fraction <30%, overt CHF, hypokalemia and alkalemia will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* serum creatinine greater then or equal to 1.5

Exclusion Criteria:

* EF<30
* Overt CHF
* Alkalemia
* Hypokalemia
* GFR<20 cc/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Incidence of contrast induced nephropathy | 48-72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jordan L Rosenstock, MD, Principal Investigator — Lenox Hill Hospital